CLINICAL TRIAL: NCT01870063
Title: Comparision of FIBTEM and Blood-loss
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Arndt-H. Kiessling, Head cardiovacular research, Johann Wolfgang Goethe University Hospital
Other Study IDs: BLUTROT
Record Dates: First submitted 2013-06-03; First posted 2013-06-05 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Sternotomy; Bleeding Test
Keywords: 5 minute bleeding test; swamb; fibtem; extem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- open heart surgery

SUMMARY:
Correlation between FIBTEM and intraoperative blood loss

ELIGIBILITY:
Inclusion Criteria:

full sternotomy age >18 Inform consent signed

Exclusion Criteria:

Hypofibrinogen

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with full sternotomy
Sampling Method: Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
bleeding | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Goethe University Hospital, Frankfurt am Main, Hesse, Germany